CLINICAL TRIAL: NCT01235845
Title: A Phase I/II Clinical Trial Evaluating DC Activated Cytokine-induced Killer Cell(DCIK) Combined With DC Treatment for Glioma
Brief Title: Dendritic Cell (DC) Activated Cytokine-induced Killer Cell (DCIK) Combined With DC Treatment for Glioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Yao Weicheng, Dou Yihe, Gao Hong, Jiao Yingbin, Zhang Xuefeng, Stemcell center of the affiliated hospital of medical colledge,Qingdao university
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCCIK001
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-11

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC-DCIK (Experimental)
  Interventions: Biological: Biological: DC activated CIK combined with DC

INTERVENTIONS:
Biological: Biological: DC activated CIK combined with DC — Dendritic cells pulsed With tumor lysate were injected back into the patient intradermally close to a lymph node, DC vaccinations will be given every week for a total of four vaccinations.
  DC activated CIK combined with IL-2 were injected intratumorally via an Ommaya reservoir every week for a total of two vaccinations.

SUMMARY:
Malignant gliomas are very aggressive and among the most common of brain tumors. A diagnosis carries with it a median survival of approximately 12 months, with 90 - 95% of patients surviving less than 2 years. The current standard treatment of surgical resection followed by radiation therapy and chemotherapy has not substantially prolonged survival.

Dendritic cells (DCs) are immune cells that form part of the mammalian immune system. Their main function is to process antigen material and present it on the surface to other cells of the immune system, thus functioning as antigen-presenting cells.In the present study, DCs were used for antigen presentation of glioma antigens to directly induce a cytotoxic T-cell response. Cytokine-induced killer (CIK)cells are shown to be a heterogeneous population, and the major population expresses both the T cell marker CD3 and the NK cell marker CD56, and is termed NKT cells, which has shown significant anti-tumor activity in both clinical trials and animal studies.

Furthermore, CIK cells are able to expand significantly when they are cultured with DCs, and the CIK cells activated by DCs stimulation (DCIKs)have a characteristic which cytotoxic activity enhanced and show increased anti-tumor activity.

This study aimed to evaluate the clinical efficacy of DCIK cells treatment combined with DCs following tumor resection and radiotherapy in patients with malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, adult patients of 18 to 70 years of age at time of diagnosis that qualify for standard treatment including surgery and radiotherapy.
2. Histologically confirmed diagnosis of 1 of the following malignant gliomas:

   Anaplastic astrocytoma Glioblastoma multiforme Oligodendroglioma Oligoastrocytoma
3. Newly diagnosed or recurrent disease
4. Patients must have had surgical resection at UCLA for the collection of their tumor. Total, subtotal, or partial resection of more then 70% of tumor mass defined by MRI.
5. After surgery, a pathological diagnosis of malignant glioma (WHO Grade III or IV) will need to be established.
6. Supratentorial tumour localisation.
7. Karnofsky performance status 60-100%
8. Life expectancy ≥ 12 weeks
9. Written informed consent of patient and/or legal guardian.
10. Must be off of steroid at least two weeks prior to vaccination
11. Hematologic and metabolic panel results will be within the parameters of the protocol.
12. Negative pregnancy test
13. Fertile patients must use effective contraception
14. Hepatitis B negative
15. Hepatitis C negative
16. HIV negative
17. Syphilis serology negative
18. Patient must have no prior sensitivity to the components of the dendritic cell vaccine.

Exclusion Criteria:

1. Anti-neoplastic chemotherapy or radiotherapy during 4 weeks before entering the study,
2. Presence of acute infection
3. Inability to obtain informed consent because of psychiatric or complicating medical problems.
4. Unstable or severe intercurrent medical or psychiatric conditions as determined by the Investigator.
5. Subjects with organ allografts.
6. Contraindication to MRI
7. Known history of autoimmune disorder
8. Subjects who have an uncontrolled systemic malignancy that is not in remission.
9. Pregnancy or breast-feeding.
10. Positive for hepatitis B, C, HIV, syphilis
11. Patients unwilling to perform a save method of birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
To assess the survival of malignant glioma | 1 year

SECONDARY OUTCOMES:
To assess the immune response of patients, to assess progression free survival and to evaluate quality of life. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Weicheng Yao, Study Chair — 2010 year
Locations (1):
- Stem cell cencter of the affiliated hospital of medical colledge,qingdao university, Qingdao, Shandong, China